CLINICAL TRIAL: NCT00802113
Title: Sequential Myeloablative Stem Cell Transplantation and Reduced Intensity Allogeneic Stem Cell Transplantation in Patients With Refractory or Recurrent Non-Hodgkin's Lymphoma and Hodgkin's Disease
Brief Title: Autologous and Allogeneic Transplant for Relapsed Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Prakash Satwani, Assistant Professor of Clinical Pediatrics, Columbia University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAA5185; CHNY-01-501 (Other: CUMC)
Record Dates: First submitted 2008-05-05; First posted 2008-12-04 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Non-Hodgkin's Lymphoma; Hodgkins Disease
Keywords: Autologous Stem Cell Transplant; Cord Blood Transplant; Allogeneic Stem Cell Transplant; Relapsed Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma | interventions — fludarabine; fludarabine phosphate; Busulfan; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - Family Donor (Experimental): Fludarabine and Busulfan: Patients who have a matched family (allogeneic) donor will go on to receive non-ablative therapy, followed by an infusion of donor stem cells; this is called an allogeneic peripheral blood stem cell transplant. The non-ablative therapy will be busulfan and ﬂudarabine, Usually large (myeloablative) doses of these drugs are used for an allogeneic transplant. However, in this study lower doses (non-ablative) of chemotherapy will be given. In patients who still have evidence of disease after allogeneic transplant, additional donor immune cells (donor lymphocyte infusion) (DLI) will be given twice to further treat the lymphoma.
  Interventions: Drug: Fludarabine; Drug: Busulfan
- Arm B - Unrelated Cord Blood or Adult (Experimental): Fludarabine, Busulfan and ATG: For patients who don't have a matched family donor, a cord blood search and unrelated adult search will be done at all of the cord blood banks and adult donor registries in the world. If a closely matched cord blood donor or unrelated adult donor is found, non-ablative chemotherapy with busulfan, ﬂudarabine and antithymocyte globulin (ATG) followed by the infusion of matched unrelated cord blood cells or adult donor stem cells or bone marrow to restore the bone marrow will be given.
  Interventions: Drug: Fludarabine; Drug: Busulfan; Drug: Anti-Thymocyte Globulin

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30 mg/m2 x 5 days
  Other Names: Fludara
Drug: Busulfan — Busulfan 3.2 mg/kg/day x 2 days
  Other Names: Busulfex
Drug: Anti-Thymocyte Globulin — Anti-Thymocyte Globulin 2.0 mg/kg/day x 4 days
  Other Names: ATG
  Arms: Arm B - Unrelated Cord Blood or Adult

SUMMARY:
The sequential combination of myeloablative therapy and autologous stem cell transplantation (APBSCT) followed by a reduced intensity allogeneic stem cell transplant (Allo SCT) and post SCT adoptive cellular immunotherapy will be well tolerated in patients with refractory or recurrent non-Hodgkin's lymphoma (NHL) and Hodgkin's disease (HD).

DETAILED DESCRIPTION:
Lymphomas are the third most common group of cancers in children and adolescents in the United States. While Hodgkin's Disease (HD) has been described for many years, some subtypes of the non-Hodgkin's Lymphomas (NHL) have only recently been described. Non-Hodgkin's lymphomas traditionally have been classified as low, intermediate or high grade based on their clinical aggressiveness. More recently they have been divided into two major subgroups indolent and aggressive lymphomas by the current National Cancer Institute (NCI/PDQ) reference. Among children, aggressive histologies are prevalent including small non-cleaved cell lymphoma, lymphoblastic lymphoma, and diffuse large cell lymphoma. The most common histologic classifications of childhood non-Hodgkin's lymphoma over the past 30 years has included the morphological schema developed by Rappaport, the morphologically and immunologically based schema of Lukes and Collins, the Kiel classifications, the prognostic sub-groupings of the National Cancer Institute's Working Formulation, and the most recently developed classification that utilizes morphological, immunophenotypic and genetic information in the Revised European-American Lymphoma (REAL) classification.

ELIGIBILITY:
Inclusion Criteria:

Patient must have adequate organ function as below

* Adequate renal function defined as:

  1. Serum creatinine less than or equal to 2.0 x normal, or
  2. Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 40 ml/min/m2 or >60 ml/min/1.73 m2 or an equivalent GFR as determined by the institutional normal range
* Adequate liver function defined as:

  1. Total bilirubin <2.0 x normal; or
  2. Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase (AST)) or serum glutamic-pyruvic transaminase (SPGT) (alanine aminotransferase (ALT)) <5.0 x normal
* Adequate cardiac function defined as:

  1. Shortening fraction of >27% by echocardiogram, or
  2. Ejection fraction of >47% by radionuclide angiogram or echocardiogram
* Adequate pulmonary function defined as:

  1. Diffusing capacity of the lungs for carbon monoxide (DLCO) >50% by pulmonary function test for autologous transplant
  2. DLCO > 40% by pulmonary function test for reduced intensity allogeneic transplant
  3. For children who are uncooperative, no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry >94% in room air.

Disease Status (Eligibility)

* Patients with Non-Hodgkin's Lymphoma with either of the following:

  1. Primary induction failure (failure to achieve initial CR) who have a partial response (PR) or stable disease (SD) with reinduction chemotherapy. *All patients are required to have a biopsy regardless of positron emission tomography (PET)/Gallium results.
  2. Patients with 1st PR, 2nd CR, 2nd PR, or 2nd SD following reinduction chemotherapy
  3. Patients with 3rd CR, 3rd PR, 3rd SD following reinduction chemotherapy
* Patients with Hodgkin's Disease with either of the following:

  1. Primary induction failure (failure to achieve initial CR) and/or primary refractory disease.
  2. First relapse

     1. Early relapse (within 12 months off therapy) (excluding those who received no therapy or radiation therapy only for initial therapy)
     2. Late relapse (greater than 12 months off therapy). Only patients with recurrent Stage III or IV disease and/or those with B symptoms at relapse (all other late relapses are excluded).
     3. Second relapse.
     4. Third relapse.
* Patients must achieve a CR, PR or SD after reinduction chemotherapy.

Exclusion Criteria:

* Patients with NHL or HD with 4th or greater CR, PR, and/or SD
* Patients with progressive disease (PD) unresponsive to reinduction chemo, radio, or immunotherapy
* Hodgkin's Disease in late relapse (other than those discussed above).
* Patients with post-transplant lymphoproliferative disease following a solid organ transplantation or AIDS associated NHL
* Patients who don't have an eligible donor
* Women who are pregnant

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2003-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Satwani, MD, Principal Investigator — Columbia University
Locations (6):
- United States (6):
  - Children's Memorial Hospital in Chicago, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - New York Medical College, Valhalla, New York
  - Duke University, Durham, North Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 30 enrolled subjects, only 23 subjects received both MAC and AutoSCT and Reduced Intensity Conditioning (RIC) and allogeneic hematopoietic cell transplantation (AlloHCT). 7 subjects did not complete the transplantation and therefore were not included into data analysis.
Groups:
- Arm A - Family Donor: Fludarabine and Busulfan: Patients who have a matched family (allogeneic) donor will go on to receive non-ablative therapy, followed by an infusion of donor stem cells; this is called an allogeneic peripheral blood stem cell transplant.
- Arm B - Unrelated Cord Blood or Adult: Fludarabine, Busulfan and ATG: For patients who don't have a matched family donor, a cord blood search and unrelated adult search will be done at all of the cord blood banks and adult donor registries in the world.
Period: Overall Study
Arm/Group | Arm A - Family Donor | Arm B - Unrelated Cord Blood or Adult
Started | 6 | 17
Completed | 6 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Family Donor | Arm B - Unrelated Cord Blood or Adult | Total
Number analyzed (Participants) | 6 | 17 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 13 | 17
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 8
  Male | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Subjects With a Complete Response (CR) Following Myeloablative Conditioning (MAC) and Autologous Stem Cell Transplantation (AutoSCT)
Description: Complete Response is defined as the complete resolution of B symptoms (i.e., weight loss, night sweats and fever) and normalization of all sites of disease on the basis of physical exam, bone marrow biopsy, and imaging studies.
Time Frame: Up to 1 year post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Family Donor | Arm B - Unrelated Cord Blood or Adult
Number analyzed (Participants) | 6 | 17
Participants | 4 | 12

2. Primary Outcome: Total Number of Subjects With a Disease Relapse or Progression Following MAC AutoSCT
Description: Includes subjects with any measurable growth of disease in a previously affected site or detection of disease in a new site confirmed by biopsy.
Time Frame: Up to 1 year post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Family Donor | Arm B - Unrelated Cord Blood or Adult
Number analyzed (Participants) | 6 | 17
Participants | 1 | 3

3. Primary Outcome: Total Number of Subjects With Partial Response or Stable Disease Following MAC AutoSCT
Description: Total includes subjects with partial response and patients with stable disease, defined as <50% reduction in measurable disease or the uninterrupted persistence of B symptoms.
Time Frame: Up to 1 year post-transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Family Donor | Arm B - Unrelated Cord Blood or Adult
Number analyzed (Participants) | 6 | 17
Participants | 4 | 9

4. Secondary Outcome: Time to Neutrophil Engraftment
Description: Following MAC AutoSCT, the median time to neutrophil (PMN) recovery will be measured.
Time Frame: Up to 1 year post-transplantation
Measure: Mean (Full Range); unit: days
Arm/Group | Arm A - Family Donor | Arm B - Unrelated Cord Blood or Adult
Number analyzed (Participants) | 6 | 17
days | 16 [14 to 18] | 24 [14 to 45]

5. Secondary Outcome: Time to Platelet Engraftment
Description: Following MAC AutoSCT, the median time to platelet recovery will be measured.
Time Frame: Up to 1 year post-transplantation
Population: 1 subject under Arm A and 2 subject under Arm B did not have this data point collected and therefore 3 subjects were not included into analysis.
Measure: Mean (Full Range); unit: days
Arm/Group | Arm A - Family Donor | Arm B - Unrelated Cord Blood or Adult
Number analyzed (Participants) | 5 | 15
days | 22 [17 to 29] | 53 [3 to 159]

6. Secondary Outcome: Total Number of Subjects With Grade II-IV Acute Graft-versus-Host-Disease (GVHD)
Description: The criteria for grading is based on extent of organ involvement (i.e., Skin, Liver and Gut - rash on >50% of skin, bilirubin 2-3 mg/dl, diarrhea > 500 ml/day) with Grade II being better outcome and Grade IV being worse outcome.
Time Frame: Up to 1 year post-transplantation
Population: Subjects who completed RIC AlloHCT
Measure: Number; unit: participants
Arm/Group | Arm A - Family Donor | Arm B - Unrelated Cord Blood or Adult
Number analyzed (Participants) | 6 | 17
participants | 0 | 7

7. Secondary Outcome: Total Number of Subjects That Experienced Transplant-related Mortality (TRM)
Description: Status as subjects died post-AlloHCT
Time Frame: Up to 1 year post-transplantation
Measure: Number; unit: participants
Arm/Group | Arm A - Family Donor | Arm B - Unrelated Cord Blood or Adult
Number analyzed (Participants) | 6 | 17
participants | 2 | 6

ADVERSE EVENTS:
Arm/Group | Arm A - Family Donor | Arm B - Unrelated Cord Blood or Adult
All-Cause Mortality (participants affected / at risk) | 2/6 | 6/17
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/17
Other Adverse Events (participants affected / at risk) | 0/6 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes